CLINICAL TRIAL: NCT06987032
Title: Improving the Hemodynamic Profile Of Chronic Renal Patients by Use of Bioimpedance
Brief Title: Hemodynamics in Chronic Kidney Disease
Acronym: HORUZ
Status: Completed | Type: Observational
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Other Study IDs: ctu2019039
Record Dates: First submitted 2025-03-21; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2021-01

CONDITIONS: Chronic Kidney Failure
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the role of thoracic and whole body bioimpedance in the hemodynamic profile of patients with chronic kidney disease.

The main question it aims to answer is:

- Is bioimpedance-determined fluid status associated with kidney function decline in patients with chronic kidney disease stage 3 - 5 (non dialysis).

DETAILED DESCRIPTION:
Participants will be measured during their regular visit to their treating nephrologist.

During a follow up of one year, 3 or 4 visits will be scheduled.

* Bioimpedance and blood pressure measurements will be achieved by non-invasive techniques.
* Blood sampling will as much as possible coincide with regular blood samplings for clinical purposes.
* All subjects will undergo echocardiography at baseline and after one year follow up.

ELIGIBILITY:
Inclusion Criteria:

* Prevalent non-dialysis patients with estimated glomerular filtration rate < 60 ml/min (for chronic kidney disease subjects)
* Age > 18 years
* Signed informed consent

Exclusion Criteria:

* Acute kidney injury
* estimated glomerular filtration rate < 20ml/min directly post-nephrectomy
* Clinical conditions affecting bioimpedance measurements: limb amputation, impaired skin integrity, brain stimulator, pacemaker with low threshold or unipolar pacemaker.
* Clinical conditions affecting body composition: liver cirrhosis, active infectious disease or any acute cardiovascular event (defined as cerebrovascular event, myocard infarction, heart failure) during the 3 months before screening for inclusion
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 206 patients with CKD stages 3-5 will be included from the outpatient clinic of Ziekenhuis Zuid-Oost Limburg in Genk (Belgium).
  A healthy control group for the cross-sectional part will be recruited through visitors and/or personnel of Ziekenhuis Oost-Limburg in Genk (Belgium).
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2021-01-09 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
whole body fluid status | Baseline, every 3 months during 1 year
  The primary objective is to associate the bioimpedance-determined fluid status [fluid overload versus non-fluid overload] with kidney function decline in patients with chronic kidney disease stage 3 (59-30ml/min), 4 (29-15ml/min) and 5 (< 15 ml/min).

SECONDARY OUTCOMES:
identify the clinical factors associated with fluid overload during a longitudinal follow up | Baseline, every 3 months during 1 year
  Secondary outcomes of interest are the central volume status (measured as ejection fraction in % by echocardiography and thoracic bioimpedance in Ohms in combination with photoplethysmography), the cardiac systolic and diastolic function (measured by echocardiography), cardiovascular events, hospitalizations, inflammatory- and nutrition status (by whole body bioimpedance measurements), and quality of life (by Short Form 36 questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Vandervoort, PhD, Principal Investigator — University Hasselt
Locations (1):
- Medicine and Life science, Hasselt, Belgium

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/32/NCT06987032/Prot_SAP_000.pdf